CLINICAL TRIAL: NCT04676854
Title: Restoration of Central Vision With the PRIMA System in Patients With Atrophic Age-Related Macular Degeneration
Brief Title: Restoration of Central Vision With the PRIMA System in Patients With Atrophic AMD
Acronym: PRIMAvera
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-PV-M
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRIMA Bionic Vision System (Experimental)
  Interventions: Device: PRIMA Bionic Vision System

INTERVENTIONS:
Device: PRIMA Bionic Vision System — Implantation of PRIMA, Vision training, follow up

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the PRIMA System in patients with atrophic AMD. Eligible subjects will be implanted with the PRIMA Implant. The subjects will be assessed with various visual function and functional vision tests at defined timepoints throughout the clinical investigation with the PRIMA System (Implant and Visual Processor).

ELIGIBILITY:
Inclusion Criteria:

* Is 60 years or older at the date of inclusion;
* Has a confirmed diagnosis of geographic atrophy due to AMD in both eyes;
* The study eye has best corrected visual acuity of logMAR 1.2 (20/320) or worse as measured by ETDRS test;
* Has an atrophic patch in the study eye including the fovea of at least the implant size (>4.5 mm2 and >2.4 mm in minimum diameter);
* Understands the constraints of the study and accepts to present for all scheduled follow-up visits;
* Patient signed informed consent

Exclusion Criteria:

* Has cataract in the study eye (with LOCS III scale NO, NC, C or P>1); (these patients will be asked to have cataract surgery performed prior to enrollment; all other patients will get IOL replacement during the PRIMA implantation);
* Underwent intra ocular lens implantation in the study eye within the last month ;
* Has a highly myopic study eye (>26 mm AP);
* Has a highly hyperopic study eye (<20 mm AP);
* Has no light perception in either eye;
* Has a history of documented choroidal neovascularization in either eye;
* Has any signs of exudative AMD including exudative AMD with detachment of retinal pigment epithelium in the central visual field of the study eye;
* Has an implanted telescope in one eye;
* Has a black IOL in the study eye;
* Has any disease (other than study allowed diseases) or condition that affects retinal function of the study eye or the visual system (e.g., central retinal artery/vein occlusion, end-stage diabetic retinopathy, Proliferative Diabetic Retinopathy (PDR), diabetic macular edema (DME), severe Non-Proliferative Diabetic Retinopathy (NPDR), retinal detachment, infectious or inflammatory retinal disease, severe glaucoma, optic neuropathy, etc.) ;
* Has any disease or condition that prevents adequate examination (including OCT) of the study eye including, but not limited to media opacities that cannot be resolved prior to implantation. Note, that this criterion is also important for the function of the implant;
* Has a corneal endothelial cell count of less than 1000 cells/mm² in the study eye;
* Suffers from nystagmus or other ocular motility disorders;
* Has any disease or condition that precludes the understanding or communication of the informed consent, study requirements or test protocols (e.g., deafness, severe multiple sclerosis, amyotrophic lateral sclerosis, severe neuritis, etc.);
* Has epileptic seizures;
* Has a known sensitivity to the contact materials of the implant (iridium oxide, silicon-carbide and titanium);
* Has a known allergy to anesthetic drugs;
* Presents with hypotonia in the study eye (<8 mmHg);
* Presents with hypertonia in the study eye (>23 mmHg with treatment);
* Has active cancer or a history of intraocular, optic nerve or brain cancer and metastasis;
* Is an immune-suppressed subject (e.g., due to HIV positive diagnosis, etc.);
* Is a known carrier of multi-resistant microorganisms;
* Is receiving anticoagulation therapy that cannot be adapted to allow eye surgery;
* Is participating in another investigational drug or device study that may interfere with the PRIMAvera study;
* Has a history of chronic or recurrent infection or inflammation that would preclude participation in the study;
* Has significant recurrent or chronic inflammations or infections. Specifically, patients with the following disorders are excluded:

  * Severe chronic and consuming diseases that frequently associated with infection (e.g. Crohn disease, Whipple's disease);
  * Active inflammation in the area of the eye (e.g. herpes of cornea and/or conjunctiva, recurrent blepharoconjunctivitis, hordeolum, chalazion);
* Has a severe psychological disorder;
* Does not have the mental capacity to legally sign the informed consent;
* Has severe renal, cardiac, hepatic, etc. organ diseases (ASA IV or worse);
* Has head dimensions that are incompatible with the PRIMA Glasses;
* Has a refraction of study eye higher than + 4 dpt or lower than - 4 dpt for patients with IOL (there is no refraction criteria for phakic patients, since they get an IOL during PRIMA implantation);
* Has too high and/or unrealistic expectations (e.g., believes that a benefit is guaranteed or expects normal vision after surgery).

The following additional exclusion criteria are applicable for French subjects:

* Is a protected person per French law (e.g. is under guardianship, person deprived of their liberty);
* Is not affiliated to a mandatory social security program (health insurance).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with meaningful improvement of visual acuity | 12 months
  Proportion of subjects with an improvement of visual acuity of logMAR 0.2 or more from baseline to 12 months
Serious Adverse Events | 12 months
  Number and severity of device and procedure related serious adverse events at 12 months follow-up

SECONDARY OUTCOMES:
Proportion of subjects with meaningful improvement of visual acuity | 6, 24, 36 months
  Proportion of subjects with an improvement of visual acuity of logMAR 0.2 or more at 6, 24 and 36 months compared to baseline
Improvement of visual acuity | 6, 12, 24, 36 months
  Mean improvement of visual acuity at 6, 12, 24 and 36 months compared to baseline
Quality of life measured by IVI | 6, 12, 24, 36 months
  IVI-Impact of Vision Impairment questionnaire (quality of life based on patient reported outcome of functional vision, participation in vision-related daily living activities and emotional well-being) at 6, 12, 24 and 36 months
Central visual perception | 12 months
  Central visual perception with PRIMA at 12 months compared to central visual perception at baseline
Adverse Events | 6, 12, 24, 36 months
  Number and severity of procedure and device related adverse events at 6, 12, 24 and 36 months follow-up
Change of natural visual acuity | 6, 12, 24, 36 months
  Change of natural visual acuity without the PRIMA Glasses
Proportion of compliant implantations | 4 weeks after implantation
  Number of subjects with PRIMA implant placed according protocol

CONTACTS AND LOCATIONS:
Locations (21):
- France (7):
  - Hôpital Pellegrin, Bordeaux
  - Centre hospitalier intercommunal de Créteil - Service Ophtalmologie, Créteil
  - Hôpital de la Croix-Rousse CHU de LYON, Lyon
  - Centre Monticelli Paradis, Marseille
  - CHU de Nantes, Nantes
  - Hopital des Quinze Vingts, Paris
  - Fondation Ophtalmologique A. De Rothschild, Paris
- Germany (10):
  - Universitätsklinikum Aachen, Klinik fuer Augenheilkunde, Aachen
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Augenklinik, Hamburg
  - Klinikum Ludwigshafen -Augenklinik, Ludwigshafen am Rhein
  - Universitätsklinikum Schleswig-Holstein Klinik für Augenheilkunde, Lübeck
  - Augenklinik der Ludwig-Maximilian Universität München, Munich
  - Universitäts-Augenklinik Münster, Münster
  - KNAPPSCHAFTSKLINIKUM SAAR GMBH Augenklinik Sulzbach, Sulzbach
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Università di Roma Tor Vergata - Policlinico Tor Vergata (PTV), Dipartimento di Medicina Sperimentale - Oftalmologia, Roma, Italy
- Rotterdam Eye Hospital, Rotterdam, Schiedamse Vest 160, Netherlands
- Instituto de Microcirugía Ocular de Barcelona, Barcelona, Spain
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palanker D, Le Mer Y, Mohand-Said S, Muqit M, Sahel JA. Photovoltaic Restoration of Central Vision in Atrophic Age-Related Macular Degeneration. Ophthalmology. 2020 Aug;127(8):1097-1104. doi: 10.1016/j.ophtha.2020.02.024. Epub 2020 Feb 25. PMID 32249038
- [Derived] Holz FG, Le Mer Y, Muqit MMK, Hattenbach LO, Cusumano A, Grisanti S, Kodjikian L, Pileri MA, Matonti F, Souied E, Stanzel BV, Szurman P, Weber M, Bartz-Schmidt KU, Eter N, Delyfer MN, Girmens JF, van Overdam KA, Wolf A, Hornig R, Corazzol M, Brodie F, Olmos de Koo L, Palanker D, Sahel JA. Subretinal Photovoltaic Implant to Restore Vision in Geographic Atrophy Due to AMD. N Engl J Med. 2026 Jan 15;394(3):232-242. doi: 10.1056/NEJMoa2501396. Epub 2025 Oct 20. PMID 41124203
- See also: Pixium Vision — http://www.pixium-vision.com